CLINICAL TRIAL: NCT05290896
Title: Correlations Between Lens Star Parameters and Phacoemulsification in Clinical Practice.
Brief Title: Correlations Between Lens Star and Phacoemulsification.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rc-3-29
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Cataract; Lens Diseases; Lens Opacities
Keywords: Cataract
MeSH Terms: conditions — Cataract; Lens Diseases | interventions — Phacoemulsification

STUDY DESIGN:
Intervention Model Description: Senile cataract patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lens star biometry (Other): Biometry done prior to phacoemulsification
  Interventions: Device: Phacoemulsification

INTERVENTIONS:
Device: Phacoemulsification — Phacoemulsification for senile cataract.
  Other Names: Phaco

SUMMARY:
To assess correlations between lens star biometry parameters and phacoemulsification in clinical practice.

DETAILED DESCRIPTION:
To analyze possible correlations between lens star biometry parameters and phacoemulsification in mild to moderate senile cataract.

ELIGIBILITY:
Inclusion Criteria:

* patients that will undergone phacoemulsification for their mild to moderate senile cataracts.

Exclusion Criteria:

* congenital and developmental cataract.
* cases with congenital lens anomalies as ectopia lentis and spheophakia.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between parameters measured by lens star. | Immediately before phacoemulsification surgery
  Anterior chamber depth, lens, axial length, keratometry readings and age of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelshafy, MD, Principal Investigator — Benha University; Marwa A Abdelshafy, MD, Study Director — Benha University
Locations (1):
- Ahmed Abdelshafy, Banhā, QA, Egypt

IPD SHARING:
Plan to Share IPD: Undecided